NCT number: NCT05722704

Official title: Effect of Cryotherapy on Post-endodontic Pain

ID: IRB/COD/STD/14/May-2022

Date: November 13, 2024

## Statistical Analysis:

Categorical data were presented as frequency and percentage values and were analyzed using the chi-square test. Numerical data were presented as mean, standard deviation (SD), median, and interquartile range (IQR) values. They were analyzed for normality using Shapiro-Wilk's test. Age data were normally distributed and were analyzed using one-way ANOVA followed by Tukey's post hoc test. Pain score data were non-parametric and were analyzed using Kruskal-Wallis's test followed by Dunn's post hoc test for intergroup comparisons and Friedman's test followed by Nemenyi post hoc test for intragroup comparisons. Correlations were analyzed using Spearman's rank-order correlation coefficient. The significance level was set at p<0.05 within all tests. Statistical analysis was performed with R statistical analysis software version 4.3.2 for Windows\*.